CLINICAL TRIAL: NCT04583761
Title: Tobacco and Nicotine Consumption and the Risk of Acquisition of COVID-19: A Case Control Study Among Healthcare Workers
Brief Title: Tobacco and Nicotine Consumption and the Risk of Acquisition of Coronavirus Disease 2019 (COVID-19)
Acronym: NICORISCOVID
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200663
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cases: Healthcare workers with mild symptoms of COVID-19 and a positive RT-PCR test for SARS-CoV-2
  Interventions: Behavioral: questionnaire
- controls: Healthcare workers with mild symptoms of COVID-19 and a negative RT-PCR test for SARS-CoV-2
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — Mailed structured regarding current and former tobacco consumption and use of alternative nicotine delivery systems

SUMMARY:
The purpose of this case-control study is to assess the association of the current and former consumption of tobacco and nicotine in the risk of acquisition of severe acute respiratory syndrome 2 (SARS-CoV-2). the investigators will send a structured interview by mail regarding use of tobacco and nicotine to 2500 healthcare workers (1250 cases with a positive Real Time Polymorphism Chain Reaction (RT-PCR) and 1250 controls with a negative PCR) who were tested in Paris for in March and April, 2020. OR will be estimated by conditional logistic regression modelling with matching for sex and age.

DETAILED DESCRIPTION:
The negative impact of tobacco use on lung health is widely recognized, together with poorer response to several infections. Smoking behaviour is characterized by inhalation and repetitive hand-to-mouth movements which could contribute to virus acquisition. In the context of SARS-CoV-2 outbreak, smoking appears to be associated with negative progression and adverse outcomes. On the other hand, several epidemiological studies suggest that the risk of infection with SARS-CoV-2 is significantly lower (OR 0.3) among current smokers, and this negative association remains significant after adjustment for age or occupation. An hypothesis is that the expression of the gene encoding for angiotensin II conversion enzyme-2-receptor could be down-regulated by nicotin. However several bias in these retrospective epidemiological studies limit their strength. Few informations are available among former smokers and users of alternative nicotine delivery systems.

In March 2020, at Hotel Dieu Hospital in Paris the investigators opened a center for SARS-CoV-2 screening, with nasopharyngeal swabs and RT-PCR, for healthcare workers who had symptoms compatible with SARS-CoV-2 (i.e. fever, chills, headaches, dry cough, anosmia, ageusia, diarrhea). No severe cases were tested. So far, more than 8000 healthcare workers had been tested, among which 40% were positive.

The aim of this study is to perform a case-control study in healthcare workers who underwent SARS-CoV-2 RT-PCR, in which cases are infected with a positive RT-PCR and controls are negative. Cases and controls will be matched for sex and age. In order to obtain with > 80% probability an OR < 0.6, the investigators estimated that the number of subjects to be included is 1250 cases and 1250 controls. A structured questionnaire assessing current and former tobacco consumption and alternative nicotine delivery systems will be sent by mail to cases and controls. Informed consent will be obtained by mail.

OR will be estimated by conditional logistic regression modelling with matching for sex and age.

Such a case-control study will elicit relevant information about the role of tobacco and nicotine use in the risk of acquisition of SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers with mild symptoms of COVID-19 tested with RT-PCR in nasopharyngeal swabs:

  * Cases : positive RT-PCR
  * Controls : negative RT-PCR
* Informed consent obtained by e-mail.

Exclusion Criteria:

* no available e-mail address
* age < 18
* no answer to the structured questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare workers tested for SARS-CoV-2 in Hotel Dieu Hospital in Paris in March, 2020
Sampling Method: Non-Probability Sample
Enrollment: 622 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
questionnaire to assess strength of correlation between current smoking and SARS-CoV-2 RT-PCR positivity | 30 minutes
  No intervention

SECONDARY OUTCOMES:
questionnaire to assess strength of correlation between current alternative nicotine delivery systems and SARS-CoV-2 RT-PCR positivity | 30 minutes
  No intervention
questionnaire to assess strength of correlation between former smokers and SARS-CoV-2 RT-PCR positivity | 30 minutes
  No intervention
questionnaire to assess strength of correlation between former alternative nicotine delivery systems and SARS-CoV-2 RT-PCR positivity | 30 minutes
  No intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel-Dieu Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No